CLINICAL TRIAL: NCT03328377
Title: The Association Between the Gut Microbiota Composition and Development of Delirium in ICU Patients
Brief Title: The Gut Microbiota and Delirium in the ICU
Acronym: GuMDel-ICU
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Herlev Hospital (Other)
Collaborators: University of Arkansas (Other)
Responsible Party: Principal Investigator, Anne Sofie Andreasen, MD, ph.d, EDIC, MD,PhD, Herlev Hospital
Other Study IDs: GuMDel-ICU
Record Dates: First submitted 2017-10-28; First posted 2017-11-01 (Actual); Last update posted 2017-11-01 (Actual); Status verified 2017-10

CONDITIONS: Delirium of Mixed Origin; Microbial Colonization
MeSH Terms: conditions — Delirium; Communicable Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Fecalsamples/Rectal swaps
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Metagenomic analysis of gut microbiota — All patients have rectal swaps/fecal samples subjected to metagenomic analysis

SUMMARY:
To investigate whether the composition of the gut microbiota is different in patients that develop delirium during critical illness as compared to patients who do not.

DETAILED DESCRIPTION:
We plan to include an equal number of patients admitted to the ICU, that either do or don't develop delirium during their course of critical illness. Samples of feces/rectal swaps will be taken at admission and again either when the patients become CAM-ICU positive, alternatively after 5 days admssion/at discharge in patients that remain CAM-ICU negative.

Samples are then sent to analyses for purification of bacterial DNA and metagenomic analysis.

ELIGIBILITY:
Inclusion Criteria: Admission to the ICU, Disability to make informed consent due to critical illness -

Exclusion Criteria: Dementia. Delirium diagnosed prior to the ICU admission on the non-ICU floors. Coma. Indication for deep sedation (-4/-5).

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Approximately 40 ICU patients and 10 healthy volunteers as controls
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2017-11-01 (Estimated); Primary Completion 2018-02-28 (Estimated); Study Completion 2018-05-31 (Estimated)

PRIMARY OUTCOMES:
Gut Microbiota composition | May 2018
  Metagenomic analysis of Gut Microbiota / composition by different bacterial families

IPD SHARING:
Plan to Share IPD: No